CLINICAL TRIAL: NCT02498678
Title: Effect of Tetanus on Neuromuscular Junction Monitor Performance in Pediatric Patients Undergoing Abdominal and / or Perineal Surgical Procedures With Using of Rocuronium
Brief Title: Effect of Tetanus on Neuromuscular Junction Monitor Performance in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ricardo Vieira Carlos, Staff Physician, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22225014.7.0000.0068
Record Dates: First submitted 2015-02-11; First posted 2015-07-15 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): After verifying the absence of sevoflurane through the gas analyzer, TOF monitor mode starts with stimuli every 12 to 15 seconds. After 1 minute (min) stimulation, calibration and supramaximal stimulation will be ensured by the built-in calibration function (CAL 2) of the TOF-Watch®. The stability of the response will be documented by at least 2 to 5 min [< 5% variation in the first response (T1) in the TOF]. Monitoring of neuromuscular junction will be held until recovery of the TOF ratio to 0.9 (90%), an expected average of 60 minutes.
- tetanus group (Experimental): After verifying the absence of sevoflurane through the gas analyzer, a 50-Hz tetanic stimulation will be applied for 5 s and followed after 1 min by TOF stimulation every 15 s. After 1 minute (min) calibration and supramaximal stimulation will be ensured by the built-in calibration function (CAL 2) of the TOF-Watch®. The stability of the response will be documented by at least 2 to 5 min [< 5% variation in the first response (T1) in the TOF]. Monitoring of neuromuscular junction will be held until recovery of the TOF ratio to 0.9 (90%), an expected average of 60 minutes.
  Interventions: Procedure: Tetanus

INTERVENTIONS:
Procedure: Tetanus — tetanic electric stimulation
  Arms: tetanus group

SUMMARY:
The objective of this study is to assess the performance of acceleromyography as a method of evaluation of muscle relaxation after application of tetanus stimulation to obtain stability of responses before administration of neuromuscular blocking agents.

DETAILED DESCRIPTION:
Effect of tetanus on neuromuscular junction monitor performance in pediatric patients undergoing abdominal and / or perineal surgical procedures with the use of rocuronium.

Routine monitoring of neuromuscular function during anesthesia offers some advantages. It helps promote proper relaxation according to each patient's individual sensitivity and reduces the possibility of postoperative residual block with its serious consequences, namely: reducing pulmonary forced vital capacity, decreased ability to increase ventilation during periods of hypoxia, increased risk of pulmonary aspiration due to lower strength of pharyngeal muscles. It can also reduce the waste of time caused by excessive paralysis. Furthermore, the interpretation of data from the monitor may indicate that pharmacological reversal of neuromuscular blockade is not required, with potential benefits over costs, as well as lower incidence of postoperative nausea and vomiting.

Acceleromyography was introduced for use in daily clinical practice in 1988 as a simple, reliable and easy to apply in the anesthetized patient monitor to assess muscle relaxation. The purpose of this neuromuscular junction (NMJ) monitor was replace mechanomyography, this modality that has greater complexity of assembling and using. The mechanomyography was considered long, the ideal objective neuromuscular monitoring. This measures the strength of isometric contraction of a muscle or digit (e.g. thumb) in response to nerve stimulation. Moreover, it requires an assembly that demands time and with strict rules for the positioning and application of non elastic preload on the thumb. This makes the method impractical for everyday use. Furthermore, monitors based on the method of mechanomyography are no longer commercially available. Acceleromyography gradually replaced mechanomyography as a method to monitor muscle relaxation in clinical practice and research.

Acceleromyography measures the acceleration (isotonic contraction) of a muscle or finger. The method is based on Newton's second law, which states that force is equal to the product of mass and acceleration. If the mass (e.g. thumb) is constant, the acceleration is directly proportional to the force. This means, in principle, it measures the unrestricted movement of the muscle in question.

Monitoring must present a stable response (baseline) for a period of 2 to 5 minutes before administration of neuromuscular blocker. The time required to reach this stable response depends on the duration of electrical stimulation and frequency in which electrical stimulation are applied. When using single mode stimulus at a frequency of 0.1 Hertz (Hz) or train-of-four (TOF) every 12 to 15 seconds, it may take 5 to 20 minutes to obtain a stable response. However, the stabilization period may be shortened by applying a short, high frequency stimulation (tetanic stimulation). Tetanic stimulation for 5 seconds can decrease the stabilization period of 2 to 5 minutes.

There is no description in the literature on the performance of tetanus stimulation in obtaining a stable response of the monitor neuromuscular junction in pediatric patients.

The objective of this study is to assess the performance of acceleromyography as a method of evaluation of muscle relaxation after application of tetanus stimulation to obtain stability of responses before administration of neuromuscular blocking agents. This performance will be compared by time of onset and recovery, recorded by the monitor during effect of neuromuscular blocking agent rocuronium; namely:

* Onset of action (height reduction of 95% in T1);
* Time to reappearance of T1, T2, T3 and T4;
* Time to TOF reaching 0.20; 0.30; 0.40; 0.50; 0.60; 0.70; 0.80; 0.90;
* Recovery interval 25-75 (elapsed time between T1 25% and T1 75%)
* Final T1 height

Materials and Methods Patient After obtaining approval by the Ethics Committee and informed consent by completing legal guardian, 50 patients (American Society of Anesthesiologists [ASA] - Physical Status 1-2, aged 2 to 11 years, regardless of genders) who will undergo abdominal and / or perineal surgery, with planned surgical time greater than 60 minutes will be included in the study. Patients with diseases or medications that are known to interfere with neuromuscular transmission, hepatic or renal dysfunction or allergy to medications used in the study will be excluded.

Anesthesia Patients will be monitored with electrocardiography, noninvasive blood pressure, pulse oximetry, capnography, gas analyzer and bispectral index. The anesthesia is induced with inhaled (sevoflurane) or intravenous (propofol and opioids) anesthetics according to the patient's ability to cooperate in obtaining venous access. The maintenance will be done with intravenous anesthesia (propofol and opioid). Peripheral temperature will be measured at the thenar eminence of the upper limb where the monitor will be installed and maintained above 32 degrees Celsius. The core temperature will be monitored in the esophagus and maintained above 35 degrees Celsius. All patients will be placed under a upper body forced air warming blanket. The trachea will be intubated without the use of muscle relaxant. Ventilation will be adjusted to maintain normocapnia (end tidal carbon dioxide 32 - 40 mmHg). Before the study began, if inhaled agents have been used for induction of anesthesia, the absence will be established by the gas analysis monitor.

Neuromuscular monitoring

Neuromuscular monitoring will follow the recommendations of good practice in research for pharmacodynamic studies of neuromuscular blocking agents. After careful cleaning of the skin, two pediatric surface electrodes will be placed in one of the upper limbs on the ulnar nerve near the wrist with a distance of 3 to 6 centimeters (cm). Upper limb and fingers will be fixed to appropriate support. The acceleromyography monitor (TOF-Watch®, Organon) will be installed on this member. Using a system of random numbers generated by computer and stored in sealed, opaque envelopes, patients will be placed in one of the following groups:

Tetanus group (n = 25) After verifying the absence of sevoflurane through the gas analyzer, a 50-Hz tetanic stimulation will be applied for 5 s and followed after 1 min by TOF stimulation every 15 s. When the response to TOF is stable, calibration and supramaximal stimulation will be ensured by the built-in calibration function (CAL 2) of the TOF-Watch®.

Control group (n = 25) After verifying the absence of sevoflurane through the gas analyzer, TOF monitor mode starts with stimuli every 12 to 15 seconds. After 1 minute (min) stimulation in the form, calibration and supramaximal stimulation will be ensured by the built-in calibration function (CAL 2) of the TOF-Watch®. If greater than 5% variation in the height of the first response (T1) of the TOF monitor will be recalibrated.

In both groups, the stability of the response will be documented by at least 2 to 5 min [<5% variation in the first response (T1) in the TOF] before administration of rocuronium.

The IV line will be inserted in the contralateral arm. The choice between the dominant and non-dominant arm will be made randomly. The dose of 0,6 milligram / kilogram of rocuronium will be administered in fast-running saline infusion within 5 seconds. The data of the TOF-Watch® monitor will be collected on a laptop using the neuromuscular junction program monitor. If needed, neuromuscular blockade will be reversed with neostigmine and atropine.

Sample Size Based on the previous study, the mean blocking time to reach TOF 0.9 is averaging 42.8 minutes, the variability from one patient to another was 9 minutes (SD = 9 minutes). (9) It is expected that, using tetanus, the average blocking time will not be less than 35 minutes on average. With 80% power and 95% confidence the sample required for conducting the study is 21 patients in each group.

Statistical Analysis Recovery times from neuromuscular blockade will be assessed between groups up to the value of TOF = 0.90. For quantitative evaluation of these parameters will be employed Student's t test or the Mann-Whitney test.

The sensitivity, parameter set automatically by the monitor, will be compared between groups. As it is also a quantitative parameter, the Student's t test or the Mann-Whitney test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Physical Status 1-2, aged 2 to 11 years, regardless of genders) who will undergo abdominal and / or perineal surgery, with planned surgical time greater than 60 minutes

Exclusion Criteria:

* Patients with diseases or medications that are known to interfere with neuromuscular transmission, hepatic or renal dysfunction or allergy to medications used in the study will be excluded

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo LA Torres, Prof., Study Director — Disciplina de Anestesiologia da FMUSP
Locations (1):
- Child Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Carlos RV, de Boer HD, Torres ML, Carmona MJ. The effect of prior tetanic stimulation on train-of-four monitoring in paediatric patients: A randomised open-label controlled trial. Eur J Anaesthesiol. 2017 Mar;34(3):163-168. doi: 10.1097/EJA.0000000000000558. PMID 27828786

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Tetanus Group
Started | 25 | 25
Completed | 25 | 23
Not Completed | 0 | 2
Not completed — interference from the surgical team | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Tetanus Group | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.8 (2.7) | 5.6 (2.35) | 6.2 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 16 | 20 | 36
Region of Enrollment [Number; unit: participants]
  Brazil | 25 | 23 | 48
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] | 17.2 (7.6) | 15.7 (1.3) | 16.5 (5.56)
Growth chart percentiles [Mean (Standard Deviation); unit: percentile] | 38.5 (27) | 44.6 (22.2) | 41.3 (24.9)
ASA physical status [Number; unit: participants] — 1. - A normal healthy patient
  2. - A patient with mild systemic disease
  participants
    1 | 15 | 18 | 33
    2 | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Train of Four 0,9 (90%)
Description: Time to recovery to train of four 0,9 (90%). When the fourth stimulus value (T4) divided by the first stimulus (T1) reaches the ratio of 0.9 (T4 / T1)
Time Frame: An expected average of 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Tetanus Group
Number analyzed (Participants) | 25 | 23
minutes | 49.9 (12.2) | 41.7 (13.1)

2. Primary Outcome: T1 Height
Description: T1 height documentation when train of four reaches 0,9 (90%)
Time Frame: An expected average of 60 minutes
Measure: Mean (Standard Deviation); unit: percentage of T1 height
Arm/Group | Control Group | Tetanus Group
Number analyzed (Participants) | 25 | 23
percentage of T1 height | 95.3 (15.8) | 69.3 (8.7)

3. Secondary Outcome: Time to Obtain T1 Height Stability
Description: Time, in minutes, for the stabilization T1 height (maximum acceptable variation of up to 5%) before administration of neuromuscular blocking agent. According to the guidelines for good clinical research practice in pharmacodynamics studies of neuromuscular blocking agents, the monitor must present a stable response of T1 height (baseline) for a period of 2-5 min before administration of an neuromuscular blocking agents.
Time Frame: An expected average of 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group | Tetanus Group
Number analyzed (Participants) | 25 | 23
seconds | 195 (203) | 116 (81.6)

4. Secondary Outcome: Monitor Settings - Electric Current
Description: Electric current (milliampere) calculated by the monitor calibration
Time Frame: An expected average of 60 minutes
Measure: Mean (Standard Deviation); unit: milliampere
Arm/Group | Control Group | Tetanus Group
Number analyzed (Participants) | 25 | 23
milliampere | 48.2 (12.1) | 47.2 (13.5)

5. Secondary Outcome: Monitor Settings - Sensitivity
Description: Sensitivity calculated by the monitor calibration, It is a numeric value that ranges from 1 to 512, but there is no measurement unit provided. Using the default CAL 2 function, the TOF-Watch® SX monitor automatically determines the sensitivity for a specific patient. The sensitivity can be adjusted between 1 and 512, where 512 represents the most sensitive setting. A sensitivity setting of 157 is the default value. This value represents how the monitor measures motor response of the patient to electrical stimulation of train of four (TOF). If the patient has intense motor response, the monitor reduces its sensitivity. If the patient has poor motor response, the monitor increase your sensitivity.
Time Frame: An expected average of 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale from 1 to 512
Arm/Group | Control Group | Tetanus Group
Number analyzed (Participants) | 25 | 23
units on a scale from 1 to 512 | 128 (41.1) | 103.8 (49.8)

ADVERSE EVENTS:
Time Frame: Reported adverse events include events starting with beginning of neuromuscular blockade monitoring and up to 24 hours after end of case
Arm/Group | Control Group | Tetanus Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No